CLINICAL TRIAL: NCT03040596
Title: The Effect of Inhaled Corticosteroids on Vocal Fold Nodules in Children: a Pilot Study
Brief Title: The Effect of Inhaled Corticosteroids on Vocal Fold Nodules in Children
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study drug no longer provided by manufacturer free of charge
Sponsor: Joseph Dohar, MD (Other)
Responsible Party: Sponsor-Investigator, Joseph Dohar, MD, Professor of Otolaryngology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY19040139
Record Dates: First submitted 2017-01-17; First posted 2017-02-02 (Estimated); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Vocal Fold Nodules
Keywords: vocal fold nodules; inhaled steroid; steroid; children; nodules
MeSH Terms: interventions — Fluticasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- inhaled steroid + voice therapy (Experimental): fluticasone inhaler, 88mcg (2 puffs), twice a day for 4 weeks + standard voice therapy
  Interventions: Drug: Fluticasone propionate; Behavioral: Standard voice therapy
- voice therapy only (Other): standard voice therapy
  Interventions: Behavioral: Standard voice therapy

INTERVENTIONS:
Drug: Fluticasone propionate — fluticasone inhaler 44mcg/puff, 2 puffs twice a day for 4 weeks
  Other Names: Flovent
  Arms: inhaled steroid + voice therapy
Behavioral: Standard voice therapy — Standard voice therapy sessions

SUMMARY:
Voice disorders are the most common communication disorder across the lifespan and vocal fold nodules are the most frequent pathology affecting voice in children. The goal of the present study is to determine the safety, feasibility, and efficacy of a short-course of inhaled corticosteroids in addition to standard voice therapy for treating vocal fold nodules.

DETAILED DESCRIPTION:
Voice disorders are the most common communication disorder across the lifespan, affecting more than 5 million school-aged children annually in the United States. Vocal fold nodules are the most frequent pathology affecting voice in children, with 21% of children negatively influenced at any given point in time, resulting in negative quality of life consequences and inferior academic performance. The traditional first-line approach to treatment of vocal fold nodules is voice therapy by Speech-Language Pathology, although corticosteroids are often implemented in conjunction with voice therapy to reduce focal inflammation at the lesion site. Operating room procedures are the traditional method to administer corticosteroids to the lesion site, although recent advances in office-based laryngeal steroid injections have become a widely popular alternative to reduce lesion size. Unfortunately, although in-office injections are more favorable to operating room procedures, due to their less invasive nature, in-office procedures are still an invasive alternative in the pediatric population. Specifically, they involve equipment that may be intimidating to the child and require the child to remain very still for prolonged periods of time, which may not be feasible with some children. Furthermore, focal vocal fold injections still involve potential adverse effects such as vocal fold hematoma. To mediate these concerns, a short course of inhaled corticosteroids may be a safe and non-invasive alternative to reducing inflammation and lesion size within the larynx. The goal of the present study is to determine the safety and feasibility of a short-course of inhaled corticosteroids in addition to standard voice therapy for treating vocal fold nodules. The study also aims to examine the effects of inhaled corticosteroids on quality of life outcomes and acoustic and aerodynamic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with vocal fold nodules;
* Considered behaviorally and cognitively appropriate by PI for voice therapy;
* English comprehension and production sufficient to participate in the protocol and in voice therapy;
* Not currently on inhaled corticosteroids;
* No previous voice therapy;
* Willing to participate in voice therapy at Children's Hospital of Pittsburgh

Exclusion Criteria:

* Other medical conditions or medications that would mask or amplify voice outcomes, including developmental or other neuromuscular conditions, major illness or disorders, chronic or acute with the exception of laryngopharyngeal reflux disease or allergies and their treatments.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
adverse events | 1 year after start of voice therapy
  number and type of adverse events
compliance with inhaler use (percent of prescribed doses marked as "taken" on diary) | 4 weeks
  percent of prescribed doses marked as "taken" on diary

SECONDARY OUTCOMES:
fundamental frequency (Hertz) | 9-12 weeks
  change in fundamental frequency from baseline to end of therapy
quality of life questionnaire | 9-12 weeks
  change in score from QOL questionnaire from baseline to end of therapy
maximum phonation time (seconds) | 9-12 weeks
  change in time from baseline to end of therapy
s/z ratio | 9-12 weeks
  change in ratio of 2 measures from baseline to end of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Dohar, MD, Principal Investigator — ENT Department, Children's Hospital of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No